CLINICAL TRIAL: NCT03081507
Title: Muslim Americans Reaching for Health and Building Alliances (MARHABA): Patient Navigation Intervention to Increase Breast and Cervical Cancer Screening Among Muslim Women in New York City
Acronym: MARHABA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 16-00803
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer; Cervical Cancer
Keywords: Muslim Americans; Patient Navigation; Breast Cancer; Cervical Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: Study participants will be randomized to an LHW-led small media intervention arm (SM-LHW) or a LHW-led patient navigation plus small media intervention arm (PN-LHW) upon determination of study eligibility and informed consent procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LHW-led small media intervention arm (SM-LHW) (Experimental)
  Interventions: Behavioral: SM-LHW
- LHW-led plus small media intervention arm (PN-LHW) (Experimental)
  Interventions: Behavioral: PN-LHW

INTERVENTIONS:
Behavioral: SM-LHW — Will not receive additional follow-up from the LHW, but will be encouraged during the session to make an appointment with their provider to schedule a mammogram and Pap test, or to consult the MARHABA webpage for information on low-cost and culturally appropriate referral sources of screening. Individuals assigned to this arm who did not attend an educational seminar will be mailed a packet containing a palm card, brochure, and letter encouraging them to speak with their provider about breast and cervical cancer screening and/or going to the MARHABA webpage. LHWs will complete a follow-up survey with participants by phone or in-person at 4 months after baseline
  Arms: LHW-led small media intervention arm (SM-LHW)
Behavioral: PN-LHW — PNLHW participants will receive three planned contacts with LHWs that focus on navigation for obtaining mammogram and/or Pap testing.The initial contact will be made by phone and will focus on motivating participants to make an appointment with their primary care provider and/or obstetrician/gynecologist (OB/GYN), as well as provide information on low-cost or free care if necessary. The second contact will discuss the process of going to the appointment and the third contact will focus on the process of obtaining and interpreting. The second and third contacts will be either made by phone or in-person, depending on participant needs.
  Arms: LHW-led plus small media intervention arm (PN-LHW)

SUMMARY:
Studies have reported Muslims in the US and NYC face numerous language and healthcare access barriers. This is a randomized randomized controlled design will be used to test the efficacy of a Patient Navigation (PN) intervention to increase participation in breast and/or cervical cancer screening among Muslim women age 40 - 75 years living in NYC. Study participants will be randomized to an Lay Health Workers (LHW) led small media intervention arm (SM-LHW) or a LHW-led patient navigation plus small media intervention arm (PN-LHW). A specific aim of the study is to develop, implement and evaluate the efficacy of a two-arm, randomized control trial designed to increase receipt of breast and/or cervical cancer screening among Muslim women aged 40 -75 years in New York City (NYC).

DETAILED DESCRIPTION:
The goal of this study, entitled Muslim Americans Reaching for Health and Building Alliances (MARHABA), is to evaluate the effectiveness of a culturally patient navigation (PN) intervention designed for Muslim women to increase breast and cervical cancer screening participation.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Muslim
* female
* residence in a NYC borough
* self-report as having received a mammogram more than two years ago and are age 40-74 years
* self-report having received a Pap test more than three years ago and are age 40-65 years

Exclusion Criteria:

* Report a past or current diagnosis of breast or cervical cancer
* Report having had a hysterectomy
* Report having had breast reconstructive surgery

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 432 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Awareness of Pap Test | 5 Months
  Pap test awareness is a positive response to the following question: "Have you ever heard of a 'Pap test'?"
Awareness of Mammogram | 5 Months
  Awareness is a positive response to the following question: "Have you ever heard of a 'mammogram'?"
Pap test receipt | 5 Months
  Pap test receipt is defined as a positive response to "Have you ever had a 'Pap test'?" after describing the test. For "no" responses, we defined Pap test intention as a positive response to "Are you planning on obtaining a 'Pap test'?"
Mammogram test receipt | 5 Months
  Mammogram test receipt is defined as a positive response to "Have you ever had a 'Mammogram'?" after describing the test. For "no" responses, we defined Mammogram test intention as a positive response to "Are you planning on obtaining a 'Mammogram'?"

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Islam, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Wyatt LC, Chebli P, Patel S, Alam G, Naeem A, Maxwell AE, Raveis VH, Ravenell J, Kwon SC, Islam NS. A Culturally Adapted Breast and Cervical Cancer Screening Intervention Among Muslim Women in New York City: Results from the MARHABA Trial. J Cancer Educ. 2023 Apr;38(2):682-690. doi: 10.1007/s13187-022-02177-5. Epub 2022 May 19. PMID 35585475